CLINICAL TRIAL: NCT02803931
Title: Assessing the Efficacy of CardiOGoniometry (CGM) to Localise the Culprit Vessel in Mixed Vessel Disease Non-ST elevatIon Myocardial infarcTION (NSTEMI)
Acronym: COGNITION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 15/YH/0270
Record Dates: First submitted 2016-02-18; First posted 2016-06-17 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Acute Coronary Syndrome
Keywords: Cardiogoniometry; Electrocardiography
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Electrocardiography

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Cardiogoniometry (Experimental): Every patient in the study will have a cardiogoniometry recording performed by the Cardiologic Explorer whilst an inpatient on the ward. This will then be taken for interpretation to see if it indicates what vessel is the culprit causing their NSTEMI. The researcher interpreting the cardiogoniometry recording will be blind to the results of the ECG and the coronary angiography,
  Interventions: Device: Cardiogoniometry
- 12-lead ECG (Active Comparator): For every patient in the study, copies of their 12-lead ECGs performed during their admission will be taken for interpretation by an independent cardiologist. This will then be taken for interpretation to see if it indicates what vessel is the culprit causing their NSTEMI.The researcher interpreting the ECG recordings will be blind to the results of the cardiogoniometry and the coronary angiography,
  Interventions: Device: 12-lead ECG

INTERVENTIONS:
Device: Cardiogoniometry — Cardiogoniometry cardiologic explorer, Enverdis GmbH medical solutions, Germany
  Arms: Cardiogoniometry
Device: 12-lead ECG
  Arms: 12-lead ECG

SUMMARY:
This study aims to test the hypothesis that cardiogoniometry (CGM) is helpful to identify the site of the culprit vessel in patients with NSTEMI in comparison to 12-lead ECG.

NSTEMI constitutes a clinical syndrome subset of acute coronary syndrome which is most usually caused by atherosclerotic coronary artery disease. It is defined by "electrocardiographic (ECG) ST-segment depression or prominent T-wave inversion and/or positive biomarkers of necrosis (e.g., troponin) in the absence of ST-segment elevation and in an appropriate clinical setting (chest discomfort or angina equivalent)". The standard 12 lead ECG is not commonly sensitive at localising the site of the culprit lesion and even coronary angiography may not always be helpful as the majority of lesions will not have angiographically evident thrombus. Patients with an ACS may have multivessel disease and it is often not possible to identify the precise site of the culprit lesion. In patients with multivessel disease, interventionists will frequently target the most severe stenosis even though this is not necessarily the acute lesion.

CGM (Cardiogoniometry cardiologic explorer, Enverdis GmbH medical solutions, Germany) is a form of 3D vector electrocardiography which can provide quantitative analysis of myocardial depolarisation and repolarisation. It has CE mark and has been shown to be more sensitive and specific than standard 12-lead ECG at diagnosing stable coronary artery disease. Furthermore, recent work has shown CGM to be more sensitive at detecting patients with NSTEMI than conventional 12-lead ECG

In summary, there is evidence that CGM is more efficacious than 12-lead ECG at the diagnosis of both stable CAD and ACS. The hope is this that the clinical application can be extended to localising ischaemia in the culprit vessel and be a valuable diagnostic aid.

The primary objective of this study is to investigate the efficacy of CGM to identify the culprit vessel in patients presenting with NSTEMI. Secondary endpoint will be to evaluate the efficacy of CGM to detect a significant coronary stenosis (defined as ≥70%) as compared to a standard 12-lead ECG

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with NSTEMI.
* Patients who have been consented to undergo coronary angiography +/- PCI as part of their routine care by their clinician.
* Aged 18 or over.
* The patient has been informed of the nature of the study and has provided full written informed consent.

Exclusion Criteria:

* Patients unable to give informed consent including those with communication difficulties due to poor English.
* Patients with on-going chest pain at rest despite medical therapy
* Patients with haemodynamic instability and / or cardiogenic shock (defined as a sustained blood pressure of <90mmHg +/- the need for inotropic support)
* Patients with STEMI
* Those unable to perform a good quality CGM: 1) Patients who are SOB at rest; 2) Patients with very frequent ectopic beat; 3) Patients in atrial fibrillation; 4) Patients with a heart rate >150 beats/min
* Patients with previous coronary artery bypass graft surgery
* Patients who are unable to receive treatment with heparin
* Patients with significant renal impairment (defined as eGFR<30ml/min)
* Females who are or could be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2016-09-06 (Actual); Study Completion 2016-09-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity of CGM | Calculated within 30 days after participant recruitment is complete.
  The sensitivity of CGM to detect the culprit vessel will be calculated.
Specificity of CGM | Calculated within 30 days after participant recruitment is complete.
  The specificity of CGM to detect the culprit vessel will be calculated.
Positive predictive value of CGM | Calculated within 30 days after participant recruitment is complete.
  The positive predictive value of CGM to detect the culprit vessel will be calculated.
Negative predicative value of CGM | Calculated within 30 days after participant recruitment is complete.
  The negative predictive value of CGM to detect the culprit vessel will be calculated.

SECONDARY OUTCOMES:
Sensitivity of ECG | Calculated within 30 days after participant recruitment is complete.
  The sensitivity of CGM to detect the culprit vessel will be calculated.
Specificity of ECG | Calculated within 30 days after participant recruitment is complete.
  The specificity of ECG to detect the culprit vessel will be calculated.
Positive predictive value of ECG | Calculated within 30 days after participant recruitment is complete.
  The positive predictive value of ECG to detect the culprit vessel will be calculated.
Negative predictive value of ECG | Calculated within 30 days after participant recruitment is complete.
  The negative predictive value of ECG to detect the culprit vessel will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Castle Hill Hospital, Hull, East Yorkshire, United Kingdom